CLINICAL TRIAL: NCT00207441
Title: Comparing ASHC and CDSMP Outcomes In Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: University of North Carolina, Chapel Hill (Other); East Carolina University (Other)
Responsible Party: Jean Goeppinger, PhD, RN, FAAN, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CDC-NCCDPHP-S2233-22/33; S2233-22/23
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Arthritis
Keywords: arthritis; chronic disease; self management; self efficacy
MeSH Terms: conditions — Arthritis; Chronic Disease

ARMS (2):
- Arthritis self management program (Experimental)
  Interventions: Behavioral: Arthritis Self management program
- Chronic Disease Self Management Program (Experimental)
  Interventions: Behavioral: Chronic Disease Self Management Program

INTERVENTIONS:
Behavioral: Arthritis Self management program
  Other Names: ASHC; AFSMP
  Arms: Arthritis self management program
Behavioral: Chronic Disease Self Management Program
  Other Names: Living Well with Chronic Conditions; Healthy Living
  Arms: Chronic Disease Self Management Program

SUMMARY:
The arthritis-specific Arthritis Self Help Course (ASHC) and the more generic Chronic Disease Self Management Program (CDSMP) teach generalizable skills for managing arthritis and other chronic diseases. In some locations it may be more feasible to combine efforts and offer the generic course rather than the arthritis-specific program. However anecdotal evidence has questioned whether people with arthritis obtain as much benefit from the more generic course as they do the arthritis-specific course. The primary purpose of this research studies is to compare health outcomes among people with arthritis who participate in either ASHC or the CDSMP. The North Carolina project is focusing primarily on African Americans from 6 rural counties in North Carolina. The results of this research will be used to guide Arthritis program recommendations on the use of ASHC and CDSMP to improve the quality of life for people with arthritis.

ELIGIBILITY:
Inclusion Criteria:

African american adults with arthritis Caucasian adults with arthritis

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 416 (Actual)
Dates: Start 2003-04; Primary Completion 2004-10 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Health related quality of life, measured at 4 and 12 months, | 4 months, 12 months
Health care utilization measured at 4 and 12 months | 4 months, 12 months

SECONDARY OUTCOMES:
Self management behaviors measured at 4 and 12 months | 4 months, 12 months
Self efficacy for arthritis management, measured at 4 and 12 months | 4 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean Goeppinger, PhD RN, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Craven County Health Department, New Bern, North Carolina, United States